CLINICAL TRIAL: NCT03267810
Title: Randomized, Double-blinded, Controlled Trial of Early-intervention TENS for the Reduction of the Prevalence and Severity of Chronic Neuropathic Pain During the First Year After Spinal Cord Injury
Brief Title: TENS Trial to Prevent Neuropathic Pain in SCI
Acronym: TENS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty with recruitment
Sponsor: University of Miami (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Elizabeth Felix, Research Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20160951; 90SI5023 (Other Grant/Funding Number: Nat. Institute on Disability, Indep. Living, and Rehab. Res.)
Record Dates: First submitted 2017-08-23; First posted 2017-08-30 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Spinal Cord Injuries
Keywords: Neuropathic Pain; Transcutaneous Electrical Nerve Stimulation
MeSH Terms: conditions — Spinal Cord Injuries; Neuralgia | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active TENS (Experimental): Participants are given 30 minutes of TENS therapy twice a week for 8 weeks.
  Interventions: Device: TENS
- Sham TENS (Sham Comparator): Electrodes are placed on participants for 30 minutes twice a week for 8 weeks without TENS stimulation.
  Interventions: Other: Sham TENS

INTERVENTIONS:
Device: TENS — TENS: TENS 7000 - : TENS applies low-level electrical current via four pads, 2 pads affixed paraspinally, at the level of the spinal cord injury, and 2 affixed on the ventral side to areas within the dermatome corresponding to the level of injury. 15 minutes of high frequency followed by 15 minutes of low frequency will be applied at each session
  Arms: Active TENS
Other: Sham TENS — Inactive electrodes - for two 15 minute trials, neither high nor low frequency.
  Arms: Sham TENS

SUMMARY:
The purpose of this research study is to: 1) test whether transcutaneous electrical nerve stimulation (TENS) after spinal cord injury can reduce the onset of post-injury neuropathic pain; and 2) to learn more about this kind of pain and who is at risk for suffering from this type of pain after spinal cord injury. Neuropathic pain is a type of pain that occurs in about 50% of people with spinal cord injury. This type of pain is usually described as "burning" or "tingling," and is present around the level of injury and/or in areas below the level of injury. The investigators' goal is to try a non-drug treatment (TENS) that may help prevent this pain from occurring. Pain symptoms will be compared between the study participants who receive active TENS and the study participants who receive a sham TENS treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18;
* Traumatic spinal cord injury;
* Date of injury occurring within four months of study enrollment.

Exclusion Criteria:

* More than four months since date of injury;
* Contraindications for the study intervention, transcutaneous electrical nerve stimulation (TENS),88 including:
* Implanted electronic device such as a pacemaker;
* Cardiovascular problems;
* Pregnancy;
* Epilepsy;
* Cancer;
* Persons with a spinal cord injury at the C2 level, as placement of TENS electrodes on the neck is not recommended;
* Cognitive dysfunction which limits the ability of the participant to adequately understand procedures and risks.
* Prisoners
* Pregnant Women

Special populations:

* Adults unable to consent: excluded from study
* Individuals -who are not yet adults: individuals who are less than 18 years old will be excluded from the study
* Pregnant women: Women who are known to be pregnant will not be recruited into the study. A pregnancy test will be administered to females prior to enrollment in TENS (or sham) treatment. Women who become pregnant before or during the 8-week TENS treatment period will be discontinued from the study. Women who become pregnant after the 8-week TENS treatment portion of the study will continue to be enrolled, and followed according to protocol guidelines (no information will be collected specifically on the pregnancy or fetus).
* Prisoners: excluded from study
* Neonates: not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Felix, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Active TENS: Participants are given 30 minutes of TENS therapy twice a week for 8 weeks.
  TENS: TENS 7000 - : TENS will apply low-level electrical current via four pads, two applied paraspinally at the level of spinal cord injury, and two applied on the ventral side of the body within the dermatome corresponding to the level of injury . 15 minutes of high frequency followed by 15 minutes of low frequency will be applied at each session
Period: Overall Study
Arm/Group | Active TENS | Sham TENS
Started | 13 | 13
Completed | 10 | 12
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Active TENS: Participants are given 30 minutes of TENS therapy twice a week for 8 weeks.
  TENS: TENS 7000 - : TENS applies low-level electrical current via four pads, 2 pads affixed paraspinally, at the level of the spinal cord injury, and 2 affixed on the ventral side to areas within the dermatome corresponding to the level of injury. 15 minutes of high frequency followed by 15 minutes of low frequency will be applied at each session
- Total: Total of all reporting groups
Arm/Group | Active TENS | Sham TENS | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] — Age in years at entry into study
  years | 33.38 (13.27) | 38.15 (17.13) | 35.77 (15.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 11 | 11 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 5 | 13
  Not Hispanic or Latino | 5 | 8 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 9 | 9 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects Who Develop Chronic Neuropathic Pain.
Description: as defined by a score of ≥2 on the Spinal Cord Injury Pain Inventory (SCIPI), a self-report scale of symptoms. SCIPI has a total score ranging from 0 to 4 with scores of >=2 screening positive for Neuropathic Pain in people with spinal cord injury
Time Frame: 12 months
Population: Analyses were performed were on all participants enrolled in each arm using the "last observation carried forward" process.
Measure: Number; unit: percentage of participants
Groups:
- Active TENS: Participants are given 30 minutes of TENS therapy twice a week for 8 weeks.
  TENS: TENS 7000 - : TENS will apply low-level electrical current via four pads affixed to the lower back area. 15 minutes of high frequency followed by 15 minutes of low frequency will be applied at each session
Arm/Group | Active TENS | Sham TENS
Number analyzed (Participants) | 13 | 13
percentage of participants | 31 | 46

2. Primary Outcome: Neuropathic Pain Symptom Inventory (NPSI) Scores
Description: NPSI has a total score ranging from 0 to 100 with the higher score indicating more severe symptoms of neuropathic pain
Time Frame: 12 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active TENS | Sham TENS
Number analyzed (Participants) | 13 | 13
score on a scale | 23 [0 to 33] | 14 [0 to 23]

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants reporting adverse events related to study treatment as evaluated by physician
Time Frame: 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Sham TENS: Electrodes are placed on participants for 30 minutes twice a week for 8 weeks without TENS stimulation.
  Sham TENS: Inactive electrodes - for two 15 minute trials
Arm/Group | Active TENS | Sham TENS
Number analyzed (Participants) | 13 | 13
Participants | 1 | 2

4. Secondary Outcome: Pain Interference With Function
Description: Self-report composite rating scale of interference of pain with activities, mood, and sleep. This scale has a total score ranging from 0 to 30, with a higher score indicating greater pain interference.
Time Frame: 12 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active TENS | Sham TENS
Number analyzed (Participants) | 13 | 13
score on a scale | 0 [0 to 11] | 1 [0 to 10]

5. Secondary Outcome: Depressive Symptoms
Description: Patient Health Questionnaire - 9 (PHQ-9) has a total score ranging from 0 to 27, with a higher score indicating greater depressive symptoms
Time Frame: 12 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active TENS | Sham TENS
Number analyzed (Participants) | 13 | 13
score on a scale | 4 [3 to 8] | 1 [1 to 5]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Active TENS | Sham TENS
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 4/13 | 4/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active TENS (N=13) | Sham TENS (N=13)
episode of severe nerve pain (General disorders) | 0 | 1
broken foot (Injury, poisoning and procedural complications) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
increased pain (General disorders) | 1 | 1
prolonged dysesthesia (General disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-18): https://cdn.clinicaltrials.gov/large-docs/10/NCT03267810/Prot_SAP_001.pdf